CLINICAL TRIAL: NCT00679562
Title: Skin Irritation : Prophetic Patch Test of Lactacyd Radiance
Brief Title: Lactacyd Radiance (Lactic Acid) Prophetic Patch Test
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_03648
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Hygiene
MeSH Terms: interventions — Lactic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Lactic Acid
- 2 (Placebo Comparator)
  Interventions: Other: Distilled water

INTERVENTIONS:
Drug: Lactic Acid — Application of occlusive patches containing test product. For 24 hours and repeat 2 weeks later for participants with no reaction to Lactacyd Radiance
  Other Names: Lactacyd Radiance
  Arms: 1
Other: Distilled water — Application of patches containing distilled water for 24 hours
  Arms: 2

SUMMARY:
Primay objective:

To evaluate the potential of the products in eliciting adverse skin reaction.

ELIGIBILITY:
Inclusion Criteria:

* Test area should have a healthy or normal skin
* Individuals free of any systemic or dermatological disorder which, in the opinion of the investigative personnel would interfere with the study results or increase the risk of adverse reaction
* Not currently use of steroid or any medication during the test

Exclusion Criteria:

* History of Allergy or Allergic Reaction to:

  * Hey Fever
  * Asthma
  * Poison Ivy
  * Food
  * Cosmetics
  * Soap
  * Detergent
  * Metal
  * Jewelry
  * Lather
  * Fabric
  * Medication

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2008-03; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Reaction after patch removal. | at 15-30 minutes and day 3

CONTACTS AND LOCATIONS:
Overall Officials: Taweeporn NATESUMROENG, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bangkok, Thailand